CLINICAL TRIAL: NCT03147248
Title: A Randomized, Parallel-Group, Phase I/III Study to Evaluate Efficacy, Pharmacokinetics and Safety Between Subcutaneous CT-P13 and Intravenous CT-P13 in Patients With Active Rheumatoid Arthritis
Brief Title: A Phase I/III Study to Evaluate Efficacy, PK and Safety Between CT-P13 SC and CT-P13 IV in Patients With Active RA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P13 3.5 (SC); 2016-002125-11 (EudraCT Number)
Record Dates: First submitted 2017-05-07; First posted 2017-05-10 (Actual); Results first posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — CT-P13; Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 was open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (6):
- Cohort 1: CT-P13 IV 3 mg/kg (Active Comparator): CT-P13 Intravenous (IV) (Infliximab), 3 mg/kg by IV infusion every 8 weeks (Part 1)
  Interventions: Biological: CT-P13
- Cohort 2: CT-P13 SC 90 mg (Experimental): CT-P13 Subcutaneous (SC) (Infliximab), 90 mg by SC injection every other week (Part 1)
  Interventions: Biological: CT-P13
- Cohort 3: CT-P13 SC 120 mg (Experimental): CT-P13 SC (Infliximab), 120 mg by SC injection every other week (Part 1)
  Interventions: Biological: CT-P13
- Cohort 4: CT-P13 SC 180 mg (Experimental): CT-P13 SC (Infliximab), 180 mg by SC injection every other week (Part 1)
  Interventions: Biological: CT-P13
- Arm 1: CT-P13 SC 120 mg (Experimental): CT-P13 SC (Infliximab), 120 mg by SC injection every other week with placebo intravenous infusion at Weeks 6, 14 and 22 (Part 2)
  Interventions: Biological: CT-P13
- Arm 2: CT-P13 IV 3 mg/kg (Active Comparator): CT-P13 IV (Infliximab), 3 mg/kg by IV infusion every 8 weeks with placebo subcutaneous injection at Week 6 and every 2 weeks thereafter up to Week 28 (Part 2)
  Interventions: Biological: CT-P13

INTERVENTIONS:
Biological: CT-P13 — CT-P13 (3 mg/kg) by IV infusion administered as a 2 hour IV infusion per dose every 8 weeks
  Other Names: Infliximab
  Arms: Cohort 1: CT-P13 IV 3 mg/kg
Biological: CT-P13 — CT-P13 (90 mg) by single SC injection every other week
  Other Names: Infliximab
  Arms: Cohort 2: CT-P13 SC 90 mg
Biological: CT-P13 — CT-P13 (120 mg) by single SC injection every other week
  Other Names: Infliximab
  Arms: Cohort 3: CT-P13 SC 120 mg
Biological: CT-P13 — CT-P13 (180 mg) by double SC 90 mg injections every other week
  Other Names: Infliximab
  Arms: Cohort 4: CT-P13 SC 180 mg
Biological: CT-P13 — CT-P13 (120 mg) by single SC injection every other week with placebo IV at Weeks 6, 14 and 22.
  Other Names: Infliximab
  Arms: Arm 1: CT-P13 SC 120 mg
Biological: CT-P13 — CT-P13 (3 mg/kg) by IV infusion administered as a 2 hour IV infusion per dose every 8 weeks with placebo SC at Week 6 and every other week thereafter up to Week 28
  Other Names: Infliximab
  Arms: Arm 2: CT-P13 IV 3 mg/kg

SUMMARY:
This is a Phase I/III Study to Evaluate Efficacy, Pharmacokinetics and Safety between CT-P13 SC and CT-P13 IV in Patients with Active Rheumatoid Arthritis (RA).

DETAILED DESCRIPTION:
A new subcutaneous infliximab formulation is developed by Celltrion, Inc. as an alternative to the intravenous regimen where subcutaneous infliximab injection typically takes less than 2 minutes. The availability of a subcutaneous formulation of infliximab would increase the treatment options available to patients, particularly those wishing to self-administer their therapy. This Phase I/III Study randomized, double-blinded (Part 2 only), multicenter, parallel-group study was designed to evaluate Efficacy, Pharmacokinetics and Safety between Subcutaneous CT-P13 and Intravenous CT-P13 in Patients with Active RA.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female between 18 and 75 years old, inclusive.
* Patient has a diagnosis of RA according to the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria for at least 6 months
* Patient has active disease as defined by the presence of 6 or more swollen joints (of 28 assessed), 6 or more tender joints (of 28 assessed) and serum C-reactive protein (CRP) concentration >0.6 mg/dL
* Patient who completed at least 3 months of treatment of oral or parenteral dosing with Methotrexate between 12.5 to 25 mg/kg (between 10 to 25 mg/week in Korea) and on stable dosing with Methotrexate for at least 4 weeks prior to the first administration of the study drug.

Exclusion Criteria:

* Patient who has previously received a biological agent for the treatment of RA and/or a TNFα inhibitor for the treatment of other disease
* Patient who has allergies to any of the excipients of infliximab or any other murine and/or human proteins or patient with a hypersensitivity to immunoglobulin product
* Patient who had current or past history of chronic infection with hepatitis C or human immunodeficiency virus (HIV)-1 or -2 or current infection with hepatitis B
* Patient who had acute infection requiring oral antibiotics within 2 weeks or parenteral injection of antibiotics within 4 weeks prior to the first administration of the study drug, other serious infection within 6 months prior to the first administration of study drug or recurrent herpes zoster or other chronic or recurrent infection within 6 weeks prior to the first administration of the study drug.
* Patient who had an indeterminate result for interferon-γ release assay (IGRA) or latent tuberculosis (TB) at Screening. For Part 2, if IGRA result was indeterminate at Screening, 1 retest was possible during the screening. If the repeated IGRA result was negative, the patient could be included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2019-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MoonSun Choi, Study Chair — Celltrion
Locations (1):
- Hanyang University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Constantin A, Caporali R, Edwards CJ, Fonseca JE, Iannone F, Keystone E, Schulze-Koops H, Kwon T, Kim S, Yoon S, Kim DH, Park G, Yoo DH. Efficacy of subcutaneous vs intravenous infliximab in rheumatoid arthritis: a post-hoc analysis of a randomized phase III trial. Rheumatology (Oxford). 2023 Aug 1;62(8):2838-2844. doi: 10.1093/rheumatology/keac689. PMID 36534825
- [Derived] Westhovens R, Wiland P, Zawadzki M, Ivanova D, Kasay AB, El-Khouri EC, Balazs E, Shevchuk S, Eliseeva L, Stanislavchuk M, Yatsyshyn R, Hrycaj P, Jaworski J, Zhdan V, Trefler J, Shesternya P, Lee SJ, Kim SH, Suh JH, Lee SG, Han NR, Yoo DH. Efficacy, pharmacokinetics and safety of subcutaneous versus intravenous CT-P13 in rheumatoid arthritis: a randomized phase I/III trial. Rheumatology (Oxford). 2021 May 14;60(5):2277-2287. doi: 10.1093/rheumatology/keaa580. PMID 33230526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from 21 study centers in 8 countries for Part 1. Participants recruited from 76 study centers (including 1 good clinical practice [GCP] noncompliant study center) in 12 countries for Part 2. The study was divided into 2 parts (Part 1 and Part 2). Thus, the patients from Part 2 were newly enrolled/randomized only for Part 2.
Pre-assignment Details: For Part 1, a total of 90 patients were screened, 50 patients were enrolled (40 screening failures) and 48 patients were randomized. For Part 2, a total of 528 patients were screened, 357 patients were enrolled and 343 patients were randomized. Of these, 5 patients from a significant GCP noncompliance site were excluded in all analysis population.
Groups:
- Cohort 1: CT-P13 IV 3 mg/kg (Part 1): Each participant received 2 CT-P13 IV infusions with a 2-week interval at Weeks 0 and 2. Then, this group received further 7 doses of CT-P13 IV 3 mg/kg (Infliximab) by IV infusion at Week 6 and every 8 weeks thereafter up to Week 54. Throughout the study, methotrexate (MTX) 12.5 to 25 mg/week (between 10 to 25 mg/week in Korea), oral and parenteral dose and folic acid (≥ 5 mg/week) were coadministered, oral dose.
- Cohort 2: CT-P13 SC 90 mg (Part 1): Each participant received 2 CT-P13 IV infusions with a 2-week interval at Weeks 0 and 2. Then, this group received CT-P13 SC 90 mg (Infliximab) by SC injection via pre-filled syringe (PFS) with a 2-week interval from Week 6. The dose of SC 90 mg was adjusted to SC 120 mg every 2 weeks after Week 30 in applicable patients in Cohort 2: CT-P13 SC 90 mg. Throughout the study, MTX 12.5 to 25 mg/week (between 10 to 25 mg/week in Korea), oral and parenteral dose and folic acid (≥ 5 mg/week) were coadministered, oral dose.
- Cohort 3: CT-P13 SC 120 mg (Part 1): Each participant received 2 CT-P13 IV infusions with a 2-week interval at Weeks 0 and 2. Then, this group received CT-P13 SC 120 mg (Infliximab) by SC injection via PFS with a 2-week interval from Week 6 up to Week 54. Throughout the study, MTX 12.5 to 25 mg/week (between 10 to 25 mg/week in Korea), oral and parenteral dose and folic acid (≥ 5 mg/week) were coadministered, oral dose.
- Cohort 4: CT-P13 SC 180 mg (Part 1): Each participant received 2 CT-P13 IV infusions with a 2-week interval at Weeks 0 and 2. Then, this group received CT-P13 SC 180 mg (Infliximab) by SC injection via PFS with a 2-week interval from Week 6. The dose of SC 180 mg was adjusted to SC 120 mg every 2 weeks after Week 30 in applicable patients in Cohort 4: CT-P13 SC 180 mg. Throughout the study, MTX 12.5 to 25 mg/week (between 10 to 25 mg/week in Korea), oral and parenteral dose and folic acid (≥ 5 mg/week) were coadministered, oral dose.
- Arm 1: CT-P13 SC 120 mg (Part 2): Each participant received 2 CT-P13 IV infusions with a 2-week interval at Weeks 0 and 2. Then, this group received CT-P13 SC 120 mg (Infliximab) by SC injection via pre-filled syringe (PFS) with a 2-week interval from Week 6 up to Week 54 with placebo IV at Weeks 6, 14, and 22. Patients in specific countries were administered CT-P13 SC via auto injector (AI) at Week 46 and every 2 weeks thereafter up to Week 54, and patients were switched back to CT-P13 SC via PFS at Week 56 and every 2 weeks thereafter up to Week 64. Throughout the study, MTX 12.5 to 25 mg/week (between 10 to 25 mg/week in Korea), oral and parenteral dose and folic acid (≥ 5 mg/week) were coadministered, oral dose.
- Arm 2: CT-P13 IV 3 mg/kg (Part 2): Each participant received 2 CT-P13 IV infusions with a 2-week interval at Weeks 0 and 2. Then, this group received CT-P13 IV 3 mg/kg (Infliximab) by IV infusion with a 8-week interval from Week 6 up to Week 22 (Weeks 6, 14 and 22) with placebo SC at Week 6 and every 2 weeks thereafter up to Week 28. CT-P13 IV were switched to receive CT-P13 SC via PFS at Week 30, and further doses with CT-P13 SC were given up to Week 54. Patients in specific countries were administered CT-P13 SC via AI at Week 46 and every 2 weeks thereafter up to Week 54, and patients were switched back to CT-P13 SC via PFS at Week 56 and every 2 weeks thereafter up to Week 64. Throughout the study, MTX 12.5 to 25 mg/week (between 10 to 25 mg/week in Korea), oral and parenteral dose and folic acid (≥ 5 mg/week) were coadministered, oral dose.
Period: Overall Study
Arm/Group | Cohort 1: CT-P13 IV 3 mg/kg (Part 1) | Cohort 2: CT-P13 SC 90 mg (Part 1) | Cohort 3: CT-P13 SC 120 mg (Part 1) | Cohort 4: CT-P13 SC 180 mg (Part 1) | Arm 1: CT-P13 SC 120 mg (Part 2) | Arm 2: CT-P13 IV 3 mg/kg (Part 2)
Started | 13 (This cohort is only for Part 1.) | 11 (This cohort is only for Part 1.) | 12 (This cohort is only for Part 1.) | 12 (This cohort is only for Part 1.) | 167 (This arm is for Part 2. All of the participants in Part 2 were screened only for Part 2.) | 176 (This arm is for Part 2. All of the participants in Part 2 were screened only for Part 2.)
Completed | 12 | 9 | 10 | 10 | 141 | 145
Not Completed | 1 | 2 | 2 | 2 | 26 | 31
Not completed — Adverse Event | 0 | 2 | 2 | 2 | 6 | 11
Not completed — Disease progression | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 12 | 9
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 4
Not completed — Prolonged Dosing Interval | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All-randomized population consisted of all randomly assigned patients at Week 6, regardless of whether or not any study drug dosing was completed. All patients in the all-randomized population were analyzed according to the treatment they randomized to at Week 6.
Groups:
- Cohort 1: CT-P13 IV 3 mg/kg (Part 1): Each participant received 2 CT-P13 IV infusions with a 2-week interval at Weeks 0 and 2. Then, this group received further 7 doses of CT-P13 IV 3 mg/kg (Infliximab) by IV infusion at Week 6 and every 8 weeks thereafter up to Week 54. Throughout the study, MTX 12.5 to 25 mg/week (between 10 to 25 mg/week in Korea), oral and parenteral dose and folic acid (≥ 5 mg/week) were coadministered, oral dose.
- Arm 1: CT-P13 SC 120 mg (Part 2): Each participant received 2 CT-P13 IV infusions with a 2-week interval at Weeks 0 and 2. Then, this group received CT-P13 SC 120 mg (Infliximab) by SC injection via PFS with a 2-week interval from Week 6 up to Week 54 with placebo IV at Weeks 6, 14, and 22. Patients in specific countries were administered CT-P13 SC via AI at Week 46 and every 2 weeks thereafter up to Week 54, and patients were switched back to CT-P13 SC via PFS at Week 56 and every 2 weeks thereafter up to Week 64.
  Throughout the study, MTX 12.5 to 25 mg/week (between 10 to 25 mg/week in Korea), oral and parenteral dose and folic acid (≥ 5 mg/week) were coadministered, oral dose.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: CT-P13 IV 3 mg/kg (Part 1) | Cohort 2: CT-P13 SC 90 mg (Part 1) | Cohort 3: CT-P13 SC 120 mg (Part 1) | Cohort 4: CT-P13 SC 180 mg (Part 1) | Arm 1: CT-P13 SC 120 mg (Part 2) | Arm 2: CT-P13 IV 3 mg/kg (Part 2) | Total
Number analyzed (Participants) | 13 | 11 | 12 | 12 | 167 | 176 | 391
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Between 18 and 65 years | 12 | 9 | 10 | 10 | 148 | 147 | 336
  >=65 years | 1 | 2 | 2 | 2 | 19 | 28 | 54
Age, Continuous [Median (Full Range); unit: years] | 40.0 [24 to 69] | 56.0 [39 to 68] | 49.5 [30 to 65] | 51.5 [32 to 68] | 52.0 [19 to 74] | 53.0 [18 to 74] | 53.0 [18 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 9 | 9 | 130 | 139 | 307
  Male | 2 | 2 | 3 | 3 | 37 | 37 | 84
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Oriental | 0 | 0 | 1 | 1 | 1 | 2 | 5
  White/Caucasian | 13 | 11 | 11 | 11 | 145 | 151 | 342
  Other | 0 | 0 | 0 | 0 | 21 | 23 | 44
Region of Enrollment [Number; unit: participants]
  Bosnia and Herzegovina | 0 | 0 | 0 | 0 | 10 | 11 | 21
  Bulgaria | 2 | 3 | 2 | 2 | 11 | 9 | 20
  Chile | 0 | 0 | 0 | 0 | 4 | 4 | 8
  Estonia | 2 | 1 | 1 | 2 | 0 | 3 | 3
  Hungary | 1 | 0 | 0 | 0 | 6 | 6 | 12
  South Korea | 0 | 0 | 1 | 1 | 1 | 2 | 3
  Latvia | 0 | 0 | 1 | 1 | 0 | 2 | 2
  Peru | 0 | 0 | 0 | 0 | 21 | 23 | 44
  Poland | 5 | 6 | 6 | 5 | 46 | 46 | 92
  Russia | 0 | 0 | 0 | 0 | 39 | 39 | 78
  Spain | 0 | 0 | 0 | 0 | 2 | 2 | 4
  Ukraine | 3 | 1 | 1 | 1 | 27 | 29 | 56

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve (AUCτ) of Infliximab at Steady State (Part 1)
Description: For Part 1, the primary pharmacokinetic (PK) endpoint of the AUCτ (area under the concentration-time curve) at steady state between Week 22 and Week 30 was analyzed in patients who received all doses (full) of study drug up to Week 30 (prior to Week 30) in the PK population. All patients in SC cohorts were randomly assigned at Week 14 in a 1:1 ratio to either Group A or B for PK monitoring visit period (Week 22 and Week 30). Therefore, AUCτ was calculated at Week 22 for Cohort 1: CT-P13 IV 3 mg/kg, Weeks 22 and 26 for Group A of SC cohorts, and Weeks 24 and 28 for Group B of SC cohorts.
Time Frame: Weeks 22 (pre-dose to 216 hours post-dose), 24 (14 days after start of administration [SOA] at Week 22), 26 (pre-dose) and 28 (42 days after SOA at Week 22), and Week 30 (pre-dose)
Population: The PK population consisted of the all-randomized population who received at least 1 full dose of study drug at Week 6 or thereafter and who had at least 1 PK concentration result after Week 6 treatment. Among them, patients who had AUCτ result at steady state were included for the primary analysis.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 1: CT-P13 IV 3 mg/kg (Part 1) | Cohort 2: CT-P13 SC 90 mg (Part 1) | Cohort 3: CT-P13 SC 120 mg (Part 1) | Cohort 4: CT-P13 SC 180 mg (Part 1)
Number analyzed (Participants) | 13 | 10 | 11 | 12
hr*ng/mL
  Week 22: number analyzed (Participants) | 13 | 5 | 5 | 6
  Week 22 | 12032957.5 (5345598.59) | 5047724.2 (2449771.86) | 7333767.0 (2765064.19) | 9930696.6 (3208367.37)
  Week 24: number analyzed (Participants) | 0 | 5 | 6 | 6
  Week 24 |  | 3272936.8 (2847811.60) | 4835631.9 (2156587.25) | 9322764.3 (2704651.44)
  Week 26: number analyzed (Participants) | 0 | 5 | 5 | 6
  Week 26 |  | 4722645.2 (2434832.19) | 7295570.5 (2261574.63) | 10402980.9 (3316415.11)
  Week 28: number analyzed (Participants) | 0 | 5 | 6 | 6
  Week 28 |  | 3231316.6 (2582286.88) | 5076458.7 (2733359.45) | 10578411.8 (3443240.82)

2. Primary Outcome: Change From Baseline of Disease Activity Score Using 28 Joint Counts (DAS28) (CRP) at Week 22 (Part 2)
Description: For Part 2, the primary efficacy endpoint was to demonstrate that CT-P13 SC 120 mg is non-inferior to CT-P13 IV 3 mg/kg at Week 22, as determined by clinical response according to mean change from baseline in DAS28 (CRP) at Week 22, using Analysis of Covariance (ANCOVA). Change from baseline for ANCOVA was defined as decrease from baseline and calculated as (DAS28 [CRP] at baseline - DAS28 [CRP] at Week 22). DAS28 (CRP) was calculated using the following formula: DAS28 (CRP) equals(=) (0.56 multiplied by [*] the square root [√] of TJC28 [tender joint count]) plus (+) (0.28 * √ of SJC28 [swollen joint count]) + (0.36 * the natural logarithm [ln](CRP [mg/L] + 1)) + (0.014 * patient global disease activity [GH] on visual analogue assessment [VAS]) + 0.96. DAS28 (CRP) provides a number on a scale from 0 to 10 indicating the current activity of patients with RA. DAS28 (CRP) score above 5.1 indicates high disease activity, whereas DAS28 (CRP) score below 3.2 indicates low disease activity.
Time Frame: Week 22
Population: Efficacy population consisted of all randomly assigned patients who received at least 1 full dose of study drug at Week 6 or thereafter and had at least 1 efficacy result after Week 6. Among them, patients who had DAS28 (CRP) at Week 22 were included for the analysis. All patients were analyzed according to the treatment they received.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1: CT-P13 SC 120 mg (Part 2) | Arm 2: CT-P13 IV 3 mg/kg (Part 2)
Number analyzed (Participants) | 162 | 168
score on a scale | 2.21 (0.221) | 1.94 (0.209)
Statistical Analysis 1: Comparison: Arm 1: CT-P13 SC 120 mg (Part 2) vs Arm 2: CT-P13 IV 3 mg/kg (Part 2); Primary efficacy analysis were analyzed using an ANCOVA considering the treatment as fixed effect and country, serum CRP concentration at Week 2 (≤0.6 mg/dL vs. >0.6 mg/dL), and body weight at Week 6 (≤100 kg vs. >100 kg) as covariates; Test type: Non-Inferiority — The non-inferiority was to be concluded if the lower limit of the two-sided 95% confidence interval (CI) for the difference in the mean change from baseline of DAS28 (CRP) at Week 22 was greater that the pre-specified non-inferiority margin of -0.6; Difference of Least square mean = 0.27, 95% CI 2-sided [0.02 to 0.52] — The least squares means and standard errors, estimate of treatment difference (CT-P13 SC 120 mg - CT-P13 IV 3 mg/kg), and 2-sided 95% CI obtained from the ANCOVA model

3. Secondary Outcome: Mean Actual Value of Disease Activity Score Using 28 Joint Counts (DAS28 [CRP]) (Part 2)
Description: The secondary endpoint was defined as descriptive statistics of actual value in disease activity measured by DAS28 (CRP) up to Week 54. The results up to Week 6 represented the efficacy of CT-P13 IV loading dose (3 mg/kg) regardless of randomized treatment arm (CT-P13 SC or CT-P13 IV) in both treatment arms. DAS28 (CRP) was calculated according to the following formula: DAS28 (CRP) = (0.56* √ of TJC28) + (0.28 * √ of SJC28) + (0.36 * ln(CRP [mg/L] + 1)) + (0.014 * GH on VAS) + 0.96. DAS28 (CRP) provides a number on a scale from 0 to 10 indicating the current activity of the patients with RA. DAS28 (CRP) score above 5.1 indicates high disease activity, whereas DAS28 (CRP) score below 3.2 indicates low disease activity.
Time Frame: Baseline, Week 2, Week 6, Week 14, Week 22, Week 30, and Week 54
Population: The efficacy population consisted of all randomly assigned patients who received at least 1 full dose of study drug (CT-P13 IV or CT-P13 SC) at Week 6 or thereafter, and who had at least 1 efficacy evaluation result after Week 6 and thereafter treatment. All patients in efficacy population were analyzed according to the treatment they received.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: CT-P13 SC 120 mg (Part 2) | Arm 2: CT-P13 IV 3 mg/kg (Part 2)
Number analyzed (Participants) | 165 | 174
score on a scale
  Baseline | 6.0 (0.75) | 5.9 (0.81)
  Week 2: number analyzed (Participants) | 164 | 172
  Week 2 | 4.7 (0.94) | 4.6 (1.05)
  Week 6 | 4.0 (1.20) | 4.1 (1.21)
  Week 14: number analyzed (Participants) | 164 | 172
  Week 14 | 3.5 (1.20) | 3.7 (1.25)
  Week 22: number analyzed (Participants) | 162 | 168
  Week 22 | 3.3 (1.10) | 3.5 (1.23)
  Week 30: number analyzed (Participants) | 157 | 159
  Week 30 | 3.0 (1.13) | 3.5 (1.23)
  Week 54: number analyzed (Participants) | 145 | 145
  Week 54 | 2.8 (1.14) | 2.9 (1.16)

4. Secondary Outcome: Number of Patients Achieving Clinical Response According to American College of Rheumatology 20% Response (ACR20) (Part 2)
Description: The secondary endpoint was defined as number of patients achieving clinical response according to ACR20 (20% response, defined by ACR) between CT-P13 SC and CT-P13 IV groups. The results up to Week 6 represented the efficacy of CT-P13 IV loading dose (3 mg/kg) regardless of randomized treatment arm (CT-P13 SC or CT-P13 IV).
  Responder according to the ACR20 criteria defined as, if they are fulfilled, a decrease of at least 20% in number of tender joints and swollen joints (0-28), and 20% improvement in 3 of the followings: patient assessment of pain on VAS (0-100 mm), patient global assessment of disease activity on VAS (0-100 mm) and physician global assessment of disease activity on VAS (0-100 mm), health assessment questionnaire disability index and CRP or ESR (erythrocyte sedimentation rate).
Time Frame: Week 2, Week 6, Week 14, Week 22, Week 30, and Week 54
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: CT-P13 SC 120 mg (Part 2) | Arm 2: CT-P13 IV 3 mg/kg (Part 2)
Number analyzed (Participants) | 165 | 174
Participants
  Week 2 | 63 | 57
  Week 6 | 107 | 103
  Week 14 | 124 | 130
  Week 22 | 139 | 137
  Week 30 | 142 | 133
  Week 54 | 132 | 125

5. Secondary Outcome: Observed Trough Serum Concentration (Ctrough) of Infliximab (Part 2)
Description: For evaluation of pharmacokinetics (PK), the secondary endpoint was defined as the analysis of trough concentration (concentration before the next study drug administration) of Infliximab up to Week 54. The samples were collected at Weeks 0, 2 and 6, and every 8 weeks up to Week 54. During PK monitoring visit (Weeks 22-30), samples were collected every 2 weeks according steady state PK sampling time point. All patients were randomly assigned at Week 14 in a 1:1:1:1 ratio to one of 4 groups (Groups A, B, C or D) for PK monitoring visit period. No PK results were obtained at Weeks 6 and 14 for SC group and Weeks 12, 20, 24, 26 and 28 for IV group due to 2 weeks and 8 weeks dosing interval, respectively.
Time Frame: SC group: Weeks 0, 2, 12, 20, 22, 24, 26, 28, 36, 44, and 52; IV group: Weeks 0, 2, 6, 14, 22, 36, 44, and 52
Population: The PK population consisted of all randomly assigned patients who received at least 1 full dose of study drug (CT-P13 IV, CT-P13 SC) at Week 6 or thereafter and who had at least 1 PK concentration result after Week 6 or thereafter treatment. All patients in PK population were analyzed according to the treatment they received.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Arm 1: CT-P13 SC 120 mg (Part 2) | Arm 2: CT-P13 IV 3 mg/kg (Part 2)
Number analyzed (Participants) | 166 | 174
μg/mL
  Week 0 | 15.73 (5.83) | 16.00 (5.99)
  Week 2 | 8.64 (5.97) | 8.81 (7.13)
  Week 6: number analyzed (Participants) | 0 | 172
  Week 6 |  | 1.89 (2.61)
  Week 12: number analyzed (Participants) | 165 | 0
  Week 12 | 12.33 (8.20) |
  Week 14: number analyzed (Participants) | 0 | 164
  Week 14 |  | 3.20 (11.14)
  Week 20: number analyzed (Participants) | 159 | 0
  Week 20 | 12.72 (9.13) |
  Week 22: number analyzed (Participants) | 42 | 156
  Week 22 | 13.19 (10.57) | 1.03 (1.85)
  Week 24: number analyzed (Participants) | 41 | 0
  Week 24 | 12.32 (8.55) |
  Week 26: number analyzed (Participants) | 40 | 0
  Week 26 | 10.73 (7.08) |
  Week 28: number analyzed (Participants) | 152 | 0
  Week 28 | 12.27 (9.75) |
  Week 36: number analyzed (Participants) | 156 | 150
  Week 36 | 12.20 (9.44) | 8.79 (8.63)
  Week 44: number analyzed (Participants) | 150 | 149
  Week 44 | 11.24 (8.51) | 9.97 (9.65)
  Week 52: number analyzed (Participants) | 146 | 147
  Week 52 | 10.98 (8.81) | 10.23 (10.08)

6. Secondary Outcome: Mean Actual Value in Serum CRP Concentration (Pharmacodynamic Parameter) (Part 2)
Description: For evaluation of pharmacodynamic (PD), the secondary endpoint was defined as concentration of CRP between 2 treatment groups up to Week 54. The blood samples for CRP were collected at Weeks 0, 2 and 6, and every 8 weeks up to Week 54.
  Patient who received the other treatment than that to which they were assigned at any point was defined as mis-randomized. One patient in IV group was mis-randomized and analyzed as SC group for PD analysis.
Time Frame: Baseline, Week 2, Week 6, Week 14, Week 22, Week 30, Week 38, Week 46, and Week 54
Population: The PD population consisted of all randomized population who received at least 1 full dose of study drug at Week 6 or thereafter and had at least 1 PD result (rheumatoid factor, anti-cyclic citrullinated peptide, CRP or ESR) after Week 6 treatment. All patients in PD population were analyzed according to the treatment they received.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm 1: CT-P13 SC 120 mg (Part 2) | Arm 2: CT-P13 IV 3 mg/kg (Part 2)
Number analyzed (Participants) | 168 | 175
mg/dL
  Baseline | 1.82 (2.37) | 2.23 (3.52)
  Week 2: number analyzed (Participants) | 167 | 173
  Week 2 | 0.47 (0.78) | 0.62 (1.43)
  Week 6 | 0.74 (1.38) | 0.98 (1.84)
  Week 14: number analyzed (Participants) | 166 | 173
  Week 14 | 0.81 (1.96) | 1.14 (2.53)
  Week 22: number analyzed (Participants) | 163 | 169
  Week 22 | 0.72 (1.33) | 1.16 (2.13)
  Week 30: number analyzed (Participants) | 158 | 160
  Week 30 | 0.67 (1.26) | 1.17 (2.14)
  Week 38: number analyzed (Participants) | 158 | 151
  Week 38 | 0.71 (1.28) | 1.08 (2.95)
  Week 46: number analyzed (Participants) | 151 | 148
  Week 46 | 0.60 (1.01) | 0.79 (1.47)
  Week 54: number analyzed (Participants) | 146 | 146
  Week 54 | 0.60 (1.01) | 0.78 (1.48)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were assessed from the date the informed consent form was signed until the last assessment date or End-of-Study (EOS) visit. The duration of the study was up to Week 62 for Part 1, and the study duration for Part 2 was up to Week 66 per country.
Description: Investigator was responsible for reporting all AEs that were observed during the study regardless of their relationship to study drug/clinical significance. Safety analysis was pre-specified to only report the most severe event if the same events were occurred to the same patient. All patients who received at least 1 (partial or full) dose of study drug at Week 6 or thereafter were included in safety analysis. But, for Part 2, one patient in IV group was mis-randomized and analyzed as SC group.
Arm/Group | Cohort 1: CT-P13 IV 3 mg/kg (Part 1) | Cohort 2: CT-P13 SC 90 mg (Part 1) | Cohort 3: CT-P13 SC 120 mg (Part 1) | Cohort 4: CT-P13 SC 180 mg (Part 1) | Arm 1: CT-P13 SC 120 mg (Part 2) | Arm 2: CT-P13 IV 3 mg/kg (Part 2)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11 | 0/12 | 0/12 | 1/168 | 4/175
Serious Adverse Events (participants affected / at risk) | 1/13 | 2/11 | 0/12 | 3/12 | 6/168 | 14/175
Other Adverse Events (participants affected / at risk) | 8/13 | 7/11 | 8/12 | 9/12 | 91/168 | 90/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: CT-P13 IV 3 mg/kg (Part 1) (N=13) | Cohort 2: CT-P13 SC 90 mg (Part 1) (N=11) | Cohort 3: CT-P13 SC 120 mg (Part 1) (N=12) | Cohort 4: CT-P13 SC 180 mg (Part 1) (N=12) | Arm 1: CT-P13 SC 120 mg (Part 2) (N=168) | Arm 2: CT-P13 IV 3 mg/kg (Part 2) (N=175)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hereditary haemochromatosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 — General disorders and administration site conditions
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pertussis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 — Preferred term reported as administration related reaction and occurred between start of administration and 24 hours from the end of IV infusion (including placebo for Part 2)
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Device loosening (Product Issues) | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Latent tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: CT-P13 IV 3 mg/kg (Part 1) (N=13) | Cohort 2: CT-P13 SC 90 mg (Part 1) (N=11) | Cohort 3: CT-P13 SC 120 mg (Part 1) (N=12) | Cohort 4: CT-P13 SC 180 mg (Part 1) (N=12) | Arm 1: CT-P13 SC 120 mg (Part 2) (N=168) | Arm 2: CT-P13 IV 3 mg/kg (Part 2) (N=175)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 6 | 4
Localized injection site reaction (General disorders) | 0 | 2 | 1 | 2 | 30 | 22 — General disorders and administration site conditions; preferred term reported as injection site reaction
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 7 | 4
Latent tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 8 | 10
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 1 | 7 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 2 | 9 | 13
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 0 | 9 | 9
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 3 | 13 | 16
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 2 | 9 — Infusion related reaction occurred between start of administration and 24 hours from the end of IV infusion (including placebo for Part 2)
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 8 | 11
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 3 | 7
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | 8 | 8
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 7 | 11
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 3 | 3
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 4 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 4 | 2
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0 | 2
Angular cheilitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 3
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 3
Otosalpingitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 3 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 2
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Systemic injection reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 2 | 3 — Systemic injection reaction occurred between start of administration and 24 hours from the SC injection (including placebo for Part 2)
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 3 | 2
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 3 | 3
Glucose urine (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 3
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 2 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 2
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 3 | 4
Beta-2 glycoprotein antibody positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Delayed hypersensitivity (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0 | 5 | 1 — Delayed hypersensitivity occurred after 24 hours from the study drug administration

LIMITATIONS AND CAVEATS:
Study was divided into 2 parts; Part 1 was designed to find the optimal dose of CT-P13 SC with small number of patients (~13 patients in each cohort) and Part 2 was designed to demonstrate noninferiority of CT-P13 SC with large number of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (4):
  • Study Protocol (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT03147248/Prot_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (Part 2) (2019-03-24): https://cdn.clinicaltrials.gov/large-docs/48/NCT03147248/SAP_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Addendum (Part 2) (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT03147248/SAP_002.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (Part 1) (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT03147248/SAP_003.pdf